CLINICAL TRIAL: NCT01347294
Title: Compare the Effect of Bleomycin and Tetradecyl Sodium Sulphate in the Treatment of Venous Malformations
Brief Title: Compare Two Different Sclerosing Agents in the Treatment of Venous Malformations
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Rune Andersen, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 1331TMF; TMF1331 (Other: OsloUH)
Record Dates: First submitted 2011-04-11; First posted 2011-05-04 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Venous Malformation
MeSH Terms: interventions — Bleomycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bleomycin + Fibrovein (Experimental): 1) Fibrovein 3% foamed with air 50/ 50. Total volum injected is the same as volume of malfomation. Volume of malformation estimated by contrast media injection before sclerotherapy.
  2) wait 5 minutes
  3) Bleomycin 1000 iu / ml. Injected volume same as volume of Fibrovein foam.
  Interventions: Drug: Bleomycin + Fibrovein
- Bleomycin (Active Comparator): Bleomycin 1000 iu/ ml. Total volum injected is the same as volume of malfomation. Volume of malformation estimated by contrast media injection before sclerotherapy.
  Interventions: Drug: Bleomycin
- Natrium Tetradecyl Sulphate (Fibrovein ) (Experimental): Fibrovein 3% foamed with air 50/ 50. Total volum injected is the same as volume of malfomation. Volume of malformation estimated by contrast media injection before sclerotherapy.
  Interventions: Drug: Fibrovein

INTERVENTIONS:
Drug: Bleomycin — Intralesional
  Other Names: Bleomycin Baxter
  Arms: Bleomycin
Drug: Fibrovein — Intralesional
  Other Names: Fibrovein S.T.D pharmaceutical products LTD
  Arms: Natrium Tetradecyl Sulphate (Fibrovein )
Drug: Bleomycin + Fibrovein — Intralesional
  Other Names: Bleomycin Baxter + Fibrovein pharmaceutical products
  Arms: Bleomycin + Fibrovein

SUMMARY:
The purpose of this study is to determine the effectiveness of bleomycin, fibrovein and bleomycin and fibrovein in the treatment of venous malformation.

DETAILED DESCRIPTION:
Patients with scanty symptoms from their vascular malformation can do well with conservative treatment and / or with aids and adaptations in daily life. Compression therapy (elastic stockings), pain medication and good counseling is adequate for many. Patients with significant symptoms, however, may require more invasive treatment. Previously, it was common with surgical removal, but serious sequelae and frequent recurrence after surgery resulted in caution. Today it is more common with intervention radiology treatment with injection of sclerosing agents into existing malformation. This type of therapy almost always requires repeated treatment sequences, sometimes over several months. Treatment aims to seal blood vessels in the malformation and / or make the patient as possible symptoms. Recurrence occurs frequently and there are many who are not completely free from symptoms. Many patients have chronic problems with pain, wounds, bleeding and / or they have a cosmetically disfiguring condition. Predicting the performance of a specific type of treatment can be very difficult.

Until now, there are some studies that have considered the effect of bleomycin / pingyangmycin (China) and ethanol in the treatment of vascular malformations. To our knowledge there is no prospective or retrospective studies that compare the efficacy and side effects of bleomycin and sodium tetradecyl sulfate (Fibrovein ™) in the treatment of VM.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Venous malformation
* Must be able to fill in questionary form
* Must be able to sign informed consent form

Exclusion Criteria:

* Kidney disease
* Lung disease
* Pregnancy or not willing to safe contraception
* Allergy to Bleomycin or Fibrovein

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Intesity, frequency and type of pain. | 1 year
  Pain will be measured before, during and after treatment. It will be asked about type, characteristics and intensity of pain. Using the Visual Analog Score 0-10, 0 beingno pain,10 being maximum pain, will be used in this matter.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Abildgaard, Phd, Study Director — Oslo Universitetssykehus, Rikshospitalet
Locations (1):
- Oslo Universitetssykehus Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No